CLINICAL TRIAL: NCT06635538
Title: One-Shot Ovarian Stimulation Protocol: A Pilot Study Investigating the Endocrine Profile
Brief Title: One-shot Ovarian Stimulation Protocol (One-shot)
Acronym: One-shot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSD-ONE-2024-09
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corifollitropin alfa (CFA) 150 mcg + Clomiphene Citrate (CC) 100 mg/day from D1 (Experimental)
  Interventions: Drug: Corifollitropin alfa (CFA) 150 mcg + Clomiphene Citrate (CC) 100 mg/day from D1; Drug: Clomiphene Citrate (CC) 100 mg/day from D1; Diagnostic Test: Monitoring cycle

INTERVENTIONS:
Drug: Corifollitropin alfa (CFA) 150 mcg + Clomiphene Citrate (CC) 100 mg/day from D1 — On day 2 or 3 of the menstrual cycle or after 5 days of pill-free interval, a single injection of 150 mcg of CFA (Stimulation Day 1) will be administered.
Drug: Clomiphene Citrate (CC) 100 mg/day from D1 — On day 2 or 3 of the menstrual cycle or after 5 days of pill-free interval, the patients will start oral administration of Clomiphene Citrate 100/day continuing up to and including the day of ovulation triggering
Diagnostic Test: Monitoring cycle — Scan controls and blood exams will be performed on stimulation days 1, 6, 8, 10 and, according to clinical needs, until trigger day.

SUMMARY:
The current prospective observational pilot study aims to evaluate the endocrine profile of a single-injection protocol (single CFA + daily oral administration of CC).

ELIGIBILITY:
Inclusion Criteria:

Age <= 40

AMH (Anti-Mullerian Hormone) 1.2-3.5 ng/ml or AFC 7-20

No family history of hereditary or chromosomal diseases

Body mass index (BMI) 18 to 30 kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Estradiol | days 1, 6, 8, 10,the day of ovulation triggering, the day of ovulation triggering day+1 and 7 days after oocyte retrieval
  Estradiol levels
Progesterone | days 1, 6, 8, 10,the day of ovulation triggering, the day of ovulation triggering day+1 and 7 days after oocyte retrieval
  Progesterone levels
Follicle stimulating hormone (FSH) | days 1, 6, 8, 10,the day of ovulation triggering, the day of ovulation triggering day+1 and 7 days after oocyte retrieval
  FSH levels
Luteinizing hormone (LH) | days 1, 6, 8, 10,the day of ovulation triggering, the day of ovulation triggering day+1 and 7 days after oocyte retrieval
  LH levels

SECONDARY OUTCOMES:
Days of stimulation | 7 -20 days from initiation of ovarian stimulation
Number of oocytes retrieved (COCs) | 7 -20 days from initiation of ovarian stimulation
Number of MII oocytes | 7 -20 days from initiation of ovarian stimulation
Follicular Output Rate (FORT) | 7 -20 days from initiation of ovarian stimulation
  expressed as the ratio between the total number of oocytes retrieved at oocyte pick-up and the number of antral follicles available at the start of stimulation
Follicle-to-oocyte index (FOI) | 7 -20 days from initiation of ovarian stimulation
  expressed as the ratio between the total number of oocytes retrieved at oocyte pick-up and the number of antral follicles available at the start of stimulation
Cancellation rate | 7 -20 days from initiation of ovarian stimulation
Ovarian hyperstimulation syndrome (OHSS) rate | Until 15 days after punction

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD, PhD, Principal Investigator — Dexeus Fertility
Locations (3):
- Spain (3):
  - Dexeus Mujer Sabadell, Sabadell, Barcelona
  - Dexeus Mujer Sant Cugat, Sant Cugat del Vallès, Barcelona
  - Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez F, Racca A, Rodriguez I, Polyzos NP. Ovarian stimulation for oocyte donation: a systematic review and meta-analysis. Hum Reprod Update. 2021 Jun 22;27(4):673-696. doi: 10.1093/humupd/dmab008. PMID 33742206
- [Background] Martinez F, Rodriguez-Purata J, Clua E, Garcia S, Coroleu B, Polyzos N. Ovarian response in oocyte donation cycles under LH suppression with GnRH antagonist or desogestrel progestin: retrospective and comparative study. Gynecol Endocrinol. 2019 Oct;35(10):884-889. doi: 10.1080/09513590.2019.1604662. Epub 2019 May 12. PMID 31081407
- [Background] Fares FA, Suganuma N, Nishimori K, LaPolt PS, Hsueh AJ, Boime I. Design of a long-acting follitropin agonist by fusing the C-terminal sequence of the chorionic gonadotropin beta subunit to the follitropin beta subunit. Proc Natl Acad Sci U S A. 1992 May 15;89(10):4304-8. doi: 10.1073/pnas.89.10.4304. PMID 1374895
- [Background] Glasier AF, Irvine DS, Wickings EJ, Hillier SG, Baird DT. A comparison of the effects on follicular development between clomiphene citrate, its two separate isomers and spontaneous cycles. Hum Reprod. 1989 Apr;4(3):252-6. doi: 10.1093/oxfordjournals.humrep.a136882. PMID 2497133
- [Background] Practice Committee of the American Society for Reproductive Medicine. Use of clomiphene citrate in infertile women: a committee opinion. Fertil Steril. 2013 Aug;100(2):341-8. doi: 10.1016/j.fertnstert.2013.05.033. Epub 2013 Jun 27. PMID 23809505
- [Background] Kerin JF, Liu JH, Phillipou G, Yen SS. Evidence for a hypothalamic site of action of clomiphene citrate in women. J Clin Endocrinol Metab. 1985 Aug;61(2):265-8. doi: 10.1210/jcem-61-2-265. PMID 3924949
- [Background] Dickey RP, Holtkamp DE. Development, pharmacology and clinical experience with clomiphene citrate. Hum Reprod Update. 1996 Nov-Dec;2(6):483-506. doi: 10.1093/humupd/2.6.483. PMID 9111183
- [Background] Teramoto S, Kato O. Minimal ovarian stimulation with clomiphene citrate: a large-scale retrospective study. Reprod Biomed Online. 2007 Aug;15(2):134-48. doi: 10.1016/s1472-6483(10)60701-8. PMID 17697488
- [Background] Messinis IE, Templeton A. Blockage of the positive feedback effect of oestradiol during prolonged administration of clomiphene citrate to normal women. Clin Endocrinol (Oxf). 1988 Nov;29(5):509-16. doi: 10.1111/j.1365-2265.1988.tb03700.x. PMID 3150950
- [Background] Melo AS, Paula CTV, Santos TLD, Faria VAC, Rufato MAF, Barboza RP, Barreto J. Corifollitropin alpha, clomiphene citrate and dydrogesterone without daily gonadotrophin: a new option of a friendly protocol for high-responder oocyte donors. JBRA Assist Reprod. 2022 Apr 17;26(2):315-320. doi: 10.5935/1518-0557.20210082. PMID 34672261
- See also: Related Info — http://www.dexeus.com